CLINICAL TRIAL: NCT04574310
Title: Evaluation of the Implantation Rate Depending on the Air Bubble Location Through Ultrasound Into the Uterine Cavity in Pre-embryo Transfer
Brief Title: Does the Air-bubble Location Influence on the Implantation Rate
Acronym: TRANSFER
Status: Completed | Type: Observational
Sponsor: IVI Vigo (Other)
Responsible Party: Sponsor
Other Study IDs: 1607-VGO-056-EM
Record Dates: First submitted 2020-09-28; First posted 2020-10-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Embryo Disorder
Keywords: embryo; pregnancy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Frozen embryo transfer (FET): Collect retrospectively data on embryo implantation rate
  Interventions: Other: Collect retrospectively data on embryo implantation rate
- Intracytoplasmic sperm injection (ICSI): Collect retrospectively data on embryo implantation rate
- oocyte donation: Collect retrospectively data on embryo implantation rate
  Interventions: Other: Collect retrospectively data on embryo implantation rate

INTERVENTIONS:
Other: Collect retrospectively data on embryo implantation rate — Collect retrospectively data on embryo implantation rate
  Groups: Frozen embryo transfer (FET); oocyte donation

SUMMARY:
The main objective of the study is to evaluate whether there is any association between the location into the uterine cavity, where the air bubbles containing the pre-embryos were placed, and the implantation rate. Therefore, the images generated during pre-embryos transfer are available in our database and studied retrospectively.

DETAILED DESCRIPTION:
The success of a reproductive treatment is determined by three variables: the pre-embryo quality, endometrial receptiveness and pre-embryo transfer. Several previous studies show a lack of agreement concerning the greatest measurement. For instance, some of them refer to the distance between the catheter and the uterine fundus, whereas some others take as a reference the air-bubble where the pre-embryos were placed.

It is for this reason that in the present study, we aim to evaluate the air bubble location ratio into the uterine cavity with reproductive success, taking into account the different variables to reach success. That is, embryo characteristics (quality, development day) endometrium preparation (cycle type, hormone levels on day 5) and even the transfer procedure (type of catheter, blood, difficulty channeling).

It is a study that aims to collect data from January 2013 to october 2019. To this end, the images generated during pre-embryos transfer are analyzed retrospectively. Therefore, it is evaluated the existing differences on implantation rate according to air-bubble placement into uterine cavity during the transfer procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patients with normal uterine anatomy, who underwent an ultrasound guided embryo transfer.
* BMI< 30kg/m2.
* Ultrasound guided embryo transfer made by the same researcher.

Exclusion Criteria:

* Presence of uterine fibroid in the anterior uterine body that make difficult the transfer visualization.
* Asherman Syndrome.
* Adenomyosis that reduces the uterine cavity visibility.
* Difficult transfers where the use of a semi-rigid cannula sheath is needed to entry into the uterine cavity.
* Previous uterine surgery that alters its anatomy.
* Istmocele

Ages: 30 Years to 50 Years | Sex: Female
Age Groups: Adult
Study Population: IVIVigo patients with a normal uterine anatomy and a single good quality embryo to transfer at blastocyst stage, performed by the same gynaecologist using the "three-drop technique" were included. All transfer were atraumatic, without blood presence, using soft catheter and with controlled ultrasound transfer. The distance between the fundus surface and the tip of catheter, the distance between the fundus and the air bubble, the endometrial thickness and the implantation rate were recorded.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Actual)
Dates: Start 2013-09-20 (Actual); Primary Completion 2019-10-25 (Actual); Study Completion 2019-10-25 (Actual)

PRIMARY OUTCOMES:
Implantation rate | Since September 2013 October 2019
  Analyze Implantation rate in the groups

CONTACTS AND LOCATIONS:
Overall Officials: Ekin DR Muñoz, MD, Principal Investigator — IVI Vigo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friedman BE, Lathi RB, Henne MB, Fisher SL, Milki AA. The effect of air bubble position after blastocyst transfer on pregnancy rates in IVF cycles. Fertil Steril. 2011 Mar 1;95(3):944-7. doi: 10.1016/j.fertnstert.2010.07.1063. PMID 20810105